CLINICAL TRIAL: NCT02233127
Title: A Longitudinal Birth Cohort Study in Rahimyar Khan, Pakistan
Brief Title: Birth Cohort in Rahimyar Khan, Pakistan
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: March of Dimes (Other); Aga Khan University (Other)
Responsible Party: Principal Investigator, Shaun Morris, Associate Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000045918
Record Dates: First submitted 2014-08-05; First posted 2014-09-08 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Child Mortality; Child Morbidity; Child Development; Child Behaviour
Keywords: Birth cohort; Pakistan; Child mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Birth Cohort: The cohort will comprise approximately 3000 pregnant women and their unborn babies, enrolled to participate in the control arm of a cluster-randomized controlled intervention trial (NCT02130856).

SUMMARY:
In 2010, 7.6 million children under the age of five died worldwide and yet the causes of only 2.7% (0.205 million) of these deaths were medically certified. A thorough understanding of the causes of child mortality is necessary to guide research efforts aimed at tackling this important global health problem. Prospective birth cohort studies present an opportunity to examine the relationships between early-life exposures and multiple health and non-health related outcomes including death, illness, and socioeconomic factors. In this study, we will provide insight into the underlying causes of child mortality by collecting high-quality data on early-life exposures and health and non-health related outcomes in the first year of life.

DETAILED DESCRIPTION:
In 2010, 7.6 million children under the age of five died worldwide (Liu et al., 2012). Notably, the burden of under-five mortality varies dramatically by country. The majority of total child deaths in 2010 were seen in Africa (3.6 million) and southeast Asia (2.1 million deaths), compared to 0.16 million and 0.28 million under-five deaths in Europe and the Americas, respectively (Liu et al., 2012). Strikingly, nearly half of the world's under-five child deaths in 2010 could be attributed to only five countries: India, Nigeria, Democratic Republic of the Congo, Pakistan, and China (Liu et al., 2012). In Pakistan alone, over 420,000 under-five child deaths occurred in 2010 (Liu et al., 2012).

A thorough understanding of the etiology of child mortality is necessary to guide research efforts aimed at tackling this important global health problem. Importantly, in 2010, the causes of only 2.7% (0.205 million) of all deaths in children under the age of five were medically certified (Liu et al., 2012), highlighting the need to gather high-quality data on the causes of mortality.

Prospective longitudinal birth cohort studies present an opportunity to examine temporal relationships between early-life exposures (i.e. prenatal, pregnancy, and early postnatal exposures) and multiple health and non-health related outcomes including mortality, morbidity, and socioeconomic position. It is well documented that exposures that occur early in life, including genetic, environmental, socioeconomic, and lifestyle factors, may have long-lasting effects on growth, development, and health outcomes throughout an individual's entire life course (Lynch & Smith, 2005). Thus, data on exposures during pregnancy and early childhood are valuable and may provide clues to the etiology of long-term outcomes.

Additional value can be gained through cross-cohort collaborations and comparisons (Larsen et al., 2013)(Paternoster et al., 2012)(Brion et al., 2011). By pooling data from multiple cohort studies, causal inferences can be made with greater confidence. In addition, through cross-country comparisons, heterogeneity in exposures is often increased making it more likely that an association between exposure and outcome will be observed. Similarly, cross-cohort comparisons enable researchers to investigate patterns associated with health, social, and economic outcomes in distinct regions of the world. These types of analyses may provide valuable insight into the underlying causes of global health inequalities.

The objective of this study is to implement a longitudinal prospective birth cohort study in Pakistan to obtain extensive and high-quality information on early-life exposures and health and non-health related outcomes in the first year of life. Concurrent to the design and implementation of this cohort study in Pakistan, similar studies are being implemented in Kenya (Coastal Region Cohort, Lead PI: Dr. Shaun Morris), Brazil (Pelotas Cohort, Lead PIs: Dr. Pedro R.C. Hallal, Dr. Diego G. Bassani and Dr. Mariangela Silveira), and South Africa (Birth to Twenty Cohort, Lead PI: Dr. Shane Norris). The investigators of each project have communicated their intent to align study materials in an effort to increase the ease of future comparisons between findings. This study will therefore be one crucial pillar in a multi-country cross-cohort comparison and presents a unique opportunity to investigate and compare the patterns that shape health and non-health related outcomes in individuals from four distinct regions in the world.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women and their home- or facility-born live newborns that consented to participate in the control arm of the intervention trial "An integrated toolkit to save newborn lives in Pakistan" (NCT02130856) will be eligible for this study

Exclusion Criteria:

* Did not consent to participate in the control arm of "An integrated toolkit to save newborn lives in Pakistan"(NCT02130856). Since the birth cohort study has been designed to utilize a portion of the data collected in the neonatal kit trial, individuals who do not enroll in the kit study will not be eligible to participate in birth cohort study as they will not have a complete set of data.
* Failure to provide consent to enroll in this study.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will be conducted in Rahimyar Khan (RYK) in Punjab Province, Pakistan and follows a longitudinal birth cohort design that will be conducted alongside a community-based, cluster randomized intervention trial in RYK (NCT02130856). In the concurrent intervention trial, approximately 6000 pregnant women and their unborn babies will be enrolled to participate in either the control or intervention arm of the trial; approximately half of the women will be enrolled to the control arm and half will be enrolled to the intervention arm. At the time of enrolment, women in the control arm of the trial will also be asked to participate in the birth cohort study.
Sampling Method: Probability Sample
Enrollment: 2271 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07-22 (Actual); Study Completion 2016-07-22 (Actual)

PRIMARY OUTCOMES:
Mortality within the first year of life | Day 3 of life, month 6 of life, month 12 of life
  Death from any cause within the first year of life. Assessed by questionnaire.

SECONDARY OUTCOMES:
Morbidity within the first year of a child's life | Day 3 of life, month 6 of life, month 12 of life
  The most common types of illness within the first year of a child's life will be assessed by questionnaire.
Development/behaviour of children aged 6 and 12 months in RYK, Pakistan | Month 6 of life, month 12 of life
  Assessed by questionnaire (12 month by adapted BSID-III)
  .

CONTACTS AND LOCATIONS:
Overall Officials: Shaun K Morris, MD, MPH, Principal Investigator — The Hospital for Sick Children; Zulfiqar A. Bhutta, PhD, MBBS, Principal Investigator — Aga Khan University and The Hospital for Sick Children
Locations (1):
- Aga Khan University, Karachi, Pakistan

REFERENCES:
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Larsen PS, Kamper-Jorgensen M, Adamson A, Barros H, Bonde JP, Brescianini S, Brophy S, Casas M, Charles MA, Devereux G, Eggesbo M, Fantini MP, Frey U, Gehring U, Grazuleviciene R, Henriksen TB, Hertz-Picciotto I, Heude B, Hryhorczuk DO, Inskip H, Jaddoe VW, Lawlor DA, Ludvigsson J, Kelleher C, Kiess W, Koletzko B, Kuehni CE, Kull I, Kyhl HB, Magnus P, Momas I, Murray D, Pekkanen J, Polanska K, Porta D, Poulsen G, Richiardi L, Roeleveld N, Skovgaard AM, Sram RJ, Strandberg-Larsen K, Thijs C, Van Eijsden M, Wright J, Vrijheid M, Andersen AM. Pregnancy and birth cohort resources in europe: a large opportunity for aetiological child health research. Paediatr Perinat Epidemiol. 2013 Jul;27(4):393-414. doi: 10.1111/ppe.12060. PMID 23772942
- [Background] Lynch J, Smith GD. A life course approach to chronic disease epidemiology. Annu Rev Public Health. 2005;26:1-35. doi: 10.1146/annurev.publhealth.26.021304.144505. PMID 15760279
- [Background] Brion MJ, Zeegers M, Jaddoe V, Verhulst F, Tiemeier H, Lawlor DA, Smith GD. Intrauterine effects of maternal prepregnancy overweight on child cognition and behavior in 2 cohorts. Pediatrics. 2011 Jan;127(1):e202-11. doi: 10.1542/peds.2010-0651. Epub 2010 Dec 27. PMID 21187310
- [Background] Paternoster L, Standl M, Chen CM, Ramasamy A, Bonnelykke K, Duijts L, Ferreira MA, Alves AC, Thyssen JP, Albrecht E, Baurecht H, Feenstra B, Sleiman PM, Hysi P, Warrington NM, Curjuric I, Myhre R, Curtin JA, Groen-Blokhuis MM, Kerkhof M, Saaf A, Franke A, Ellinghaus D, Folster-Holst R, Dermitzakis E, Montgomery SB, Prokisch H, Heim K, Hartikainen AL, Pouta A, Pekkanen J, Blakemore AI, Buxton JL, Kaakinen M, Duffy DL, Madden PA, Heath AC, Montgomery GW, Thompson PJ, Matheson MC, Le Souef P; Australian Asthma Genetics Consortium (AAGC); St Pourcain B, Smith GD, Henderson J, Kemp JP, Timpson NJ, Deloukas P, Ring SM, Wichmann HE, Muller-Nurasyid M, Novak N, Klopp N, Rodriguez E, McArdle W, Linneberg A, Menne T, Nohr EA, Hofman A, Uitterlinden AG, van Duijn CM, Rivadeneira F, de Jongste JC, van der Valk RJ, Wjst M, Jogi R, Geller F, Boyd HA, Murray JC, Kim C, Mentch F, March M, Mangino M, Spector TD, Bataille V, Pennell CE, Holt PG, Sly P, Tiesler CM, Thiering E, Illig T, Imboden M, Nystad W, Simpson A, Hottenga JJ, Postma D, Koppelman GH, Smit HA, Soderhall C, Chawes B, Kreiner-Moller E, Bisgaard H, Melen E, Boomsma DI, Custovic A, Jacobsson B, Probst-Hensch NM, Palmer LJ, Glass D, Hakonarson H, Melbye M, Jarvis DL, Jaddoe VW, Gieger C; Genetics of Overweight Young Adults (GOYA) Consortium; Strachan DP, Martin NG, Jarvelin MR, Heinrich J, Evans DM, Weidinger S; EArly Genetics & Lifecourse Epidemiology (EAGLE) Consortium. Meta-analysis of genome-wide association studies identifies three new risk loci for atopic dermatitis. Nat Genet. 2011 Dec 25;44(2):187-92. doi: 10.1038/ng.1017. PMID 22197932